CLINICAL TRIAL: NCT05251441
Title: The Effect of Time to Start Breast Milk Fortifiers on Neonatal Outcomes in Very Low Birth Weight Premature Infants.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 26379996
Record Dates: First submitted 2021-09-24; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-09

CONDITIONS: Breast Milk Fortifier Supplements; Premature
Keywords: Breast Milk Fortifier; Nutrition
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- F50 (Experimental): Patients in the group in which fortification was started when enteral nutrition reached 50 cc/kg
  Interventions: Dietary Supplement: Breast Milk Fortifier supplements
- F100 (Active Comparator): Patients in the group in which fortification was started when enteral nutrition reached 100 cc/kg
  Interventions: Dietary Supplement: Breast Milk Fortifier supplements

INTERVENTIONS:
Dietary Supplement: Breast Milk Fortifier supplements — Current information is recommended for breast milk supplementation in premature babies. However, there is no consensus on when it will start. For breast milk supplementation, we planned to supplement one group of our patients with enteral nutrition of 50 ml/kg/day and the other group when they reached 100 ml/kg/day.
  Other Names: F50

SUMMARY:
In the study, very low birth weight babies born in our hospital will be randomized in the closed envelope method, and breast milk fortifier will be started when 50 ml/kg/day breastfeeding volume is reached in one group, and breast milk enrichment will be started when 100 ml/kg/day enteral feeding is reached in the other group. In the study, the babies in these two groups will be compared by making early (nutrition characteristics and premature morbidity) and long-term follow-ups. In this study, a 30% reduction in the transition time to full enteral nutrition between the groups corresponds to a difference of approximately 5 days. In our study, the sample size was determined as at least 78 patients in each group, with a margin of error of 0.05 and a power of 80% to show the 5-day difference between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies born weighing less than 1500 grams

Exclusion Criteria:

* Babies with congenital anomalies
* Infants who develop necrotizing enterocolitis or spontaneous intestinal perforation before starting a breast milk fortifier
* Babies lost before reaching 50 cc/kg enteral nutrition
* Babies who are not breastfed

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
The effect of time to start breast milk fortifiers on full enteral feeding day. | 1 year
  In this study, a 30% reduction in transition time to full enteral nutrition between the groups corresponds to a difference of approximately 5 days. In the study, the sample size was determined as at least 78 patients in each group, with a margin of error of 0.05 and a power of 80% to show the 5-day difference between the groups.

SECONDARY OUTCOMES:
Weight gain rate (grams/day) | 1 year
Duration of parenteral nutrition (days) | 1 year
Time to discharge (days) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah SD, Dereddy N, Jones TL, Dhanireddy R, Talati AJ. Early versus Delayed Human Milk Fortification in Very Low Birth Weight Infants-A Randomized Controlled Trial. J Pediatr. 2016 Jul;174:126-131.e1. doi: 10.1016/j.jpeds.2016.03.056. Epub 2016 Apr 23. PMID 27112041
- [Background] Basu S, Upadhyay J, Singh P, Kumar M. Early versus late fortification of breast milk in preterm infants: a systematic review and meta-analysis. Eur J Pediatr. 2020 Jul;179(7):1057-1068. doi: 10.1007/s00431-020-03677-6. Epub 2020 May 27. PMID 32458060
- [Background] Maas C, Wiechers C, Bernhard W, Poets CF, Franz AR. Early feeding of fortified breast milk and in-hospital-growth in very premature infants: a retrospective cohort analysis. BMC Pediatr. 2013 Nov 4;13:178. doi: 10.1186/1471-2431-13-178. PMID 24180239